CLINICAL TRIAL: NCT07115381
Title: A Study on the Intervention Effect of Therapeutic Horticulture Based on the Healing System on Non-suicidal Self-injury in Adolescent Patients With Depression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lei Huang (Other)
Responsible Party: Sponsor-Investigator, Lei Huang, nurse, Guangzhou Medical University
Organization: Guangzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: (2025) No. (015)
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Horticultural Therapy; Nursing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Routine treatment and nursing
  Interventions: Other: Routine treatment and nursing
- Therapeutic Horticulture group (Experimental): Routine treatment and nursing and Therapeutic Horticulture
  Interventions: Behavioral: Therapeutic Horticulture; Other: Routine treatment and nursing

INTERVENTIONS:
Behavioral: Therapeutic Horticulture — Therapeutic Horticulture uses plant cultivation and related gardening activities as the medium of action, allowing patients to participate in gardening activities such as planting, maintenance, and harvesting of plants.
  Arms: Therapeutic Horticulture group
Other: Routine treatment and nursing — The conventional treatment mainly involves the use of antidepressant drugs, supplemented by physical therapy, psychological therapy, and rehabilitation training, etc. The routine care includes admission introduction, health education (manifestations, hazards, treatment methods of depression and non-suicidal self-harm, as well as the importance of following medical advice for treatment), medication guidance, discharge guidance, and psychological care, etc.

SUMMARY:
Non-suicidal self-harm is a serious issue. Adolescents with depression are among the high-risk groups for non-suicidal self-harm behavior. Therapeutic gardening uses plant cultivation and corresponding gardening activities as the medium of action, allowing patients to obtain therapeutic benefits by participating in gardening activities such as planting, maintaining, and harvesting plants. Therefore, this study will apply therapeutic gardening based on the healing system to adolescents with depression who have non-suicidal self-harm behavior, in order to improve their non-suicidal self-harm behavior, negative emotions, emotional expression disorders, self-efficacy, sleep quality, and loneliness.

DETAILED DESCRIPTION:
Based on the theories of positive psychology and the healing system theory framework, referring to relevant domestic and foreign literature and consulting books such as "Introduction to Horticultural Therapy", "Horticultural Rehabilitation Therapy Techniques", and "Horticultural Therapy: Growing Good Health for the Body and Mind", an intervention plan was formulated under the guidance of experts. A randomized controlled trial design was adopted. It is planned to carry out therapeutic horticulture based on the healing system for adolescent patients with depression who have non-suicidal self-harming behaviors, according to the intervention plan. By evaluating and comparing the changes and differences in indicators such as non-suicidal self-harming behaviors, emotions, physical functions, skills, and social interaction of the experimental group and the control group before and after the intervention, the actual effect of therapeutic horticulture based on the healing system in reducing the occurrence of non-suicidal self-harming behaviors among adolescent patients was verified. Finally, data analysis and paper writing were conducted.

ELIGIBILITY:
Inclusion Criteria:

* It meets the diagnostic criteria for moderate to severe depression in the Fifth Edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
* It meets the diagnostic criteria for non-suicidal self-harm in the Fifth Edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
* The patients and their guardians gave informed consent and voluntarily participated in this study.
* Have normal reading comprehension ability, language communication ability and writing ability.

Exclusion Criteria:

* Include mental disorders such as mental retardation, autism spectrum disorder, stereotyped movement disorder with self-harm, etc.
* Have had or currently have central nervous system diseases, endocrine system diseases, and other serious physical disorders.
* Are currently receiving or have received any form of systematic horticultural therapy within the past 3 months.
* Have allergic reactions to pollen, soil, or other substances that may be encountered during the intervention process.
* Have a risk of suicide and suicidal behavior.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The level and frequency of non-suicidal self-injury | Day 1 and Day 14
  The adolescent self-harm questionnaire was used to measure.This questionnaire is a self-assessment form, consisting of 19 items. Among them, the frequency of non-suicidal self-injury behavior is scored using the Likert 4-point scale: "0 times" is scored 0 points, "1 time" is scored 1 point, "2-4 times" is scored 2 points, and "5 times or more" is scored 3 points. The degree of physical harm caused is scored using the Likert 5-point scale: "No" is scored 0 points, "Mild" is scored 1 point, "Moderate" is scored 2 points, "Severe" is scored 3 points, and "Extremely severe" is scored 4 points. NSSI equivalence is equal to the product of the NSSI frequency score and the NSSI severity score. The higher the score, the more severe the condition.

SECONDARY OUTCOMES:
depressive symptom | Day 1 and Day 14
  Hamilton Depression Rating Scale-17 was used to measure.There are a total of 17 items. The lowest score of the Hamilton Depression Scale - 17 items (HAMD-17) is 0, and the highest score is 52. A total score of ≥ 24 may indicate severe depression; a score of 17 ≤ total score < 24 may indicate mild or moderate depression; a total score of ≤ 7 may indicate no depression. The higher the score, the more severe the depressive symptoms.
sleep quality | Day 1 and Day 14
  The Pittsburgh Sleep Quality Index was used to measure.This scale is used to assess an individual's recent sleep quality. It consists of 19 self-assessment items and 5 other-rater items. The 19th self-assessment item and the 5 other-rater items do not contribute to the scoring. The first 18 items cover subjective sleep quality, sleep onset time, sleep duration, sleep efficiency, sleep disorders, hypnotic drugs, and daytime functional impairment. Each factor is scored on a scale of 0 to 3, and the total score of all factors is the PSQI total score. The total score ranges from 0 to 21, and a higher PSQI total score indicates poorer sleep quality.
alexithymia | Day 1 and Day 14
  The Toronto Alexithymia Scale was used to measure.The scale consists of 20 items, including three factors: inability to identify emotions, inability to describe emotions, and extroverted thinking. It uses a 5-point scale from 1 (completely disagree) to 5 (completely agree), with a total score range of 20 to 100. The higher the score, the more severe the alexithymia is.
loneliness | Day 1 and Day 14
  The UCLA loneliness Scale was used to measure.This scale is used to assess an individual's level of loneliness, consisting of 20 items, with a 4-point rating scale ranging from 1 to 4. Some of the items are reverse-scored. The total score is the sum of the scores of each item. The total score ranges from 20 to 80, with a higher total score indicating a stronger sense of loneliness.
self-efficacy | Day 1 and Day 14
  The general self-efficacy scale was used to measure.This scale consists of 10 items. It uses a 4-point rating system, where "completely incorrect" is scored as 1 point, "somewhat correct" as 2 points, "mostly correct" as 3 points, and "completely correct" as 4 points. The highest score is 40 points and the lowest score is 10 points. The higher the score, the higher the level of self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Zhichun Xia, Study Director — The Affiliated Brain Hospital of Guangzhou Medical University
Locations (1):
- The Affiliated Brain Hospital, Guangzhou Medical University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No